CLINICAL TRIAL: NCT04287244
Title: Transcutaneous Direct Current Stimulation of the Spinal Cord for Treatment of Spasticity in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Rechdi Ahdab, M.D , PhD, Clinical Professor, Lebanese American University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LAUMCRH.RA4.11/apr/2019
Record Dates: First submitted 2020-02-19; First posted 2020-02-27 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Spastic Parapareses
MeSH Terms: conditions — Paraparesis, Spastic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tSDCS (Experimental): Anodal tSDCS will be administered through a pair of conductive rubber electrodes covered by saline soaked sponges (35 cm2). The current will be delivered continuously at 2 mA for 30 min through a battery-driven constant-current stimulator (designed by Sooma). The anode will be positioned over the spinal cord area at the level of the spinous processes of 10th-11th thoracic vertebra.
  Interventions: Device: Transcutaneous Spinal Direct Current Stimulation
- Sham tSDCS (Sham Comparator): Sham stimulation will be delivered to the same spinal cord area using a sham tSDCS device that delivers a direct current for 10 seconds at the beginning and end of tSDCS to provide sensory experiences similar to active stimulation.
  Interventions: Device: Transcutaneous Spinal Direct Current Stimulation

INTERVENTIONS:
Device: Transcutaneous Spinal Direct Current Stimulation — tSDCS will be administered through a pair of conductive rubber electrodes covered by saline soaked sponges (35 cm2). The current will be delivered continuously at 2 mA for 30 min through a battery-driven constant-current stimulator (Sooma Oy, Helsinki, Finland).

SUMMARY:
The current research is aimed at using Transcutaneous Spinal Direct Current Stimulation (tSDCS) as complementary therapeutic tool in the treatment of spasticity in multiple sclerosis. Patients will be randomized into two groups (tSDCS-anode vs. tSDCS-sham) according to the detailed protocol. Main outcome will be measured by the change in walking speed using the Timed 25-Foot Walk (T25FW).

A total of 40 patients ought to be enrolled as specified in methodology. Secondary outcomes will assess functional improvement through Multiple Sclerosis Walking Scale (MSWS) Short Form - 36 (SF-36), Expanded Disability Status Scale (EDSS) and Ashworth scale.

DETAILED DESCRIPTION:
Spasticity is experienced in around 80 % of patients with multiple sclerosis resulting in quality of life impairment. Transcranial direct current stimulation has been proven effective for the treatment of spasticity in patients with chronic stroke or cerebral palsy. The effect of transcutaneous spinal direct current stimulation (tSDCS) has been applied in spasticity but not in patients with spasticity due to multiple sclerosis. The study aims to assess the efficacy of anodal tSDCS on spasticity in multiple sclerosis patients through several assessment tools. The investigators hypothesize that anodal tSDCS will reduce spasticity in multiple sclerosis patients.

The study will be double blind sham-controlled crossover. The patients will be examined by the described assessment tools (T25FW, MSWS, SF-36, Ashworth, EDSS) before receiving tSDCS. The sessions of tSDCS will be applied 1 session per day in 5 consecutive days. Assessment using the scales and questionnaires will be performed at the end of the 5 days of stimulation, 1 week after the last day of first block of sessions and 2 weeks later. The group will be crossed and another block of 5 consecutive days of stimulation will follow. Assessment will take place again on first day and last day of the stimulations followed as well by assessment 1 week after the last day of second block of stimulation and 2 weeks after.

ELIGIBILITY:
Inclusion Criteria:

-Patients diagnosed with Multiple Sclerosis according to the 2010 Mc Donald criteria with spasticity in the lower extremities

Exclusion Criteria:

* Cardiac pacemakers
* Patients with prior exposure to tDCS
* Metallic hardware in the spine
* Eczema or skin abrasion at the intended site of stimulation
* Currently pregnant or plan for pregnancy in the next 6 months
* Heart or respiratory failure resulting in activity impairment
* Walking impairment due to orthopaedics condition such as deformity or recent fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Gait improvement | 5 days
  The primary objective of the study is to achieve 20% gait speed improvement on 25 feet walking test (T25WT) after spasticity reduction by cathodal tSDCS.

SECONDARY OUTCOMES:
Spasticity Assessment | 19 days
  Assessment by Ashworth scale (0-4)
Multiple Sclerosis Walking Assessment | 19 days
  Using Multiple Sclerosis Walking Scale (0-12)
Quality of Life Measures | 19 days
  Assessed through Short Form - 36 (0-100)
Disability Measure | 19 days
  Through Extended Disability Status Scale (0-10)